CLINICAL TRIAL: NCT03619798
Title: Evaluation of HemoTypeSC as a Novel Rapid Test for Point-of-Care Screening for Sickle-Cell Disease, Hemoglobin C Disease, and Carrier Status in Low-Resource Settings: a Multi-Center
Brief Title: Evaluation of HemoTypeSC as a Novel Rapid Test for Point-of-Care Screening for Sickle-Cell Disease, Hemoglobin C Disease, and Carrier Status in Low-Resource Settings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Silver Lake Research Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HTSC111
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HemoTypeSC — Point-of-Care Rapid Test for Detection of Sickle Cell Disease-Relevant Hemoglobin Phenotypes in Whole Blood

SUMMARY:
Sickle cell disease is a life-threatening genetic disorder that can be effectively treated following early diagnosis via newborn screening. However, sickle cell disease is most prevalent in low-resource regions of the world, where newborn screening is rare due to the cost and logistical burden of laboratory-based methods. In many such regions, >80% of affected children die, undiagnosed, before the age of five years. A convenient and inexpensive point-of-care test for sickle cell disease is thus crucially needed. In this study we will conduct a blinded, multicenter, prospective diagnostic accuracy study of HemoTypeSC(TM), an inexpensive 15-minute point-of-care immunoassay for detecting sickle cell disease, hemoglobin C disease, and trait phenotypes in newborns, children, and adults.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to be enrolled (or has parent/guardian approval to be enrolled)

Exclusion Criteria:

* Previous sickle cell screening

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newborns, children, and adults from neonatal intensive care clinics, maternity wards, and other clinics at various low-, medium-, and high-resource study centers in multiple countries.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive for Hemoblogin A, S, or C | Immediate (investigational test) to one week (reference test)
Negative for Hemoglobin A, S, or C | Immediate (investigational test) to one week (reference test)
Positive for Hemoglobin AA, AS, AC, SS, SC, or CC | Immediate (investigational test) to one week (reference test)
Negative for Hemoglobin AA, AS, AC, SS, SC, or CC | Immediate (investigational test) to one week (reference test)

CONTACTS AND LOCATIONS:
Locations (1):
- Silver Lake Research Corporation, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: Undecided